CLINICAL TRIAL: NCT01549184
Title: Retrospective Analysis of the Safety and Efficacy of Hydroxychloroquine in Immune Thrombocytopenia Among 40 Patients
Brief Title: Retrospective Analysis of the Safety and Efficacy of Hydroxychloroquine in Immune Thrombocytopenia
Acronym: HCQITP
Status: Completed | Type: Observational
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Khellaf Mehdi, Principal Investigator, Henri Mondor University Hospital
Other Study IDs: HCQITP; HCQ ITP (Other: Referral center for autoimmune cytopenia among adults)
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Immune Thrombocytopenia; Systemic Lupus Erythematosus
Keywords: secondary ITP; hydroxychloroquine; Systemic Lupus Erythematosus
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospective study of the safety and efficacy of hydroxychloroquine among patients with immune Thrombopenia (ITP).

DETAILED DESCRIPTION:
Hydroxychloroquine (HCQ) is usually used in Patients with Systemic Lupus Erythematosus (SLE) in order to treat mainly arthralgia or skin manifestations of this disease. A few studies have previously shown that HCQ could also be useful for treating autoimmune cytopenia and particularly autoimmune thrombopenia associated with SLE. In this retrospective study, the investigators have selected patients followed in our center and who have received HCQ either for an authentic SLE or because they had positive antinuclear antibodies (> 1/160e on HEP2 cells) without a definite SLE according to the American College of Rheumatology.

The main goal of this study is to compare the efficacy of HCQ in these two subgroups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Immune Thrombopenia according to the American Society of Hematology (ASH) guidelines 2011
* Positive antinuclear antibodies > 1/160e on Hep2 cells

Exclusion Criteria:

* Secondary ITP (eg HIV, HCV, HBV, lymphoproliferative disorders...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients with an immune thrombopenia with or without a definite SLE have been retrospectively studied. All the patients should have an ITP according to the ASH guidelines 2011 and have positive antinuclear antibodies (title >1/160e on Hep2 cells).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving a response (Platelet count > 30x10^9/L and doubling of the baseline count) or a complete response (platelet count > 100x10^9/L for a t least 6 months) | one year
  Time to achieve a response, concomittant(s) treatment(s), need for an emergency treatment

SECONDARY OUTCOMES:
Tolerance of Hydroxychloroquine | one year
  allergy, myopathy HCQ induced

REFERENCES:
- [Derived] Khellaf M, Chabrol A, Mahevas M, Roudot-Thoraval F, Limal N, Languille L, Bierling P, Michel M, Godeau B. Hydroxychloroquine is a good second-line treatment for adults with immune thrombocytopenia and positive antinuclear antibodies. Am J Hematol. 2014 Feb;89(2):194-8. doi: 10.1002/ajh.23609. Epub 2013 Nov 20. PMID 24254965